CLINICAL TRIAL: NCT05149001
Title: Study Among People Living With HIV and Their Health Professionals of Associated Factors of Resilience to Self-stigma
Acronym: RESILSTIGMA
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Poitiers University Hospital (Other); Poissy-Saint Germain Hospital (Other); Centre Hospitalier Universitaire Dijon (Other); Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other); Hopital Antoine Beclere (Other); Nantes University Hospital (Other); Hospital, La Roche sur Yon (Unknown); Hôpital Necker-Enfants Malades (Other); Centre Hospitalier de Bretagne Sud (Other); Reims University hospital (Other); Groupe Hospitalier de la Rochelle Ré Aunis (Other); Hospital Laennec, Quimper (Unknown); University Hospital, Brest (Other); Hospital Cornouaille, Quimper (Unknown); Centre Hospitalier de Cholet (Other); University Hospital, Strasbourg (Other); CH Annecy Genevois (Other); Centre hospitalier de Perpignan (Other); Centre Hospitalier le Mans (Other); Centre Hospitalier VALENCIENNES (Other); Bicetre Hospital (Other); Centre Hospitalier Universitaire de Nice (Other); University Hospital, Marseille (Other); Jacques Lacarin Hospital Center (Other); L'hôpital Nord-Ouest - Villefranche Villefranche sur Saône (Other); Centre Hospitalier Universitaire de Besancon (Other); Hospital, Vannes (Unknown); Moulins Hospital (Other); Hospital, Montluçon (Unknown); Centre Hospitalier de Niort (Other); Hôpital Edouard Herriot (Other); Hospital La Source, Orléans (Unknown); Centre Hospitalier du Pays d'Aix (Other); Hospital Andre Mignot, Le Chesnay (Unknown); Hôpital Raymond Poincaré (Other); University Hospital, Angers (Other Government); University Hospital, Pointe-à-Pitre (Unknown); Centre Hospitalier des Pays de Morlaix (Other); Hospital Foch, Suresnes (Unknown); Tenon Hospital, Paris (Other); University Hospital of Saint-Etienne (Other); Centre Hospitalier de Saint-Denis (Other); University Hospital, Mulhouse (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 JACOMET 2; 2021-A01588-33 (Other: ANSM)
Record Dates: First submitted 2021-11-29; First posted 2021-12-08 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2021-11

CONDITIONS: HIV Infections
Keywords: HIV; Stigmatization; Self-stigma
MeSH Terms: conditions — HIV Infections; Stereotyping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is perform to study the effect of psychological and psychosocial factors associated with resilience to the self-stigmatization of people living with HIV

DETAILED DESCRIPTION:
Epidemiological and sociological survey carried out with patients and their caregivers in the CHUs and CHGs of France via the COREVIH from 01/17/2022 to 02/17/2022.

Primary endpoint: Self-stigmatization as experienced by PLWHA will be explored through a patient questionnaire Secondary endpoints:The main explanatory variables will be studied by means of a custom questionnaire intended for the patient and covering psychological flexibility, social provisions, avoidance and fusion mechanisms, quality of life, anxiety and depression.

The socio-demographic explanatory variables will be collected by questionnaire, covering the following areas: sex, age, geographical origin, insecurity, drug use, sexuality, family context, employment, leisure, care environment.

A questionnaire intended for caregivers will study the self-stigmatization perception of the people they care for and the means implemented to fight against self-stigmatization.

Anonymous data will be reported in Redcap. The population will be described by numbers and percentages for categorical variables and by the mean ± standard deviation or the median [interquartile range] for the quantitative variables, with regard to their statistical distribution. Normality will be studied by the Shapiro-Wilk test and / or by histogram. As far as possible, graphical representations will be associated with the analyzes.

ELIGIBILITY:
Inclusion Criteria:

* For patients: adult patient, male or female, infected with HIV medically monitored in a hospital department involved in the investigation.
* Affiliation to a Social Security scheme For caregivers:Caregiver caring for people living with HIV as part of a hospital service involved in the survey (doctor, IDE, psychologist, other ...).

Exclusion Criteria:

* Minor patient
* Refusal of participation
* Persons under guardianship, guardianship or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people living with HIV
Sampling Method: Probability Sample
Enrollment: 667 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Self-stigma as experienced by PLHIV will be explored through a custom questionnaire intended for the patient | 1 day during the scheduled consultation in the infectious diseases department of the Gabriel Montpied University Hospital in Clermont-Ferrand
  Percentage of patient with self-stigma

SECONDARY OUTCOMES:
The main explanatory variables will be studied by means of a custom questionnaire intended for the patient | 1 day during the scheduled consultation in the infectious diseases department of the Gabriel Montpied University Hospital in Clermont-Ferrand
  multivariate analysis of factors associated with disparition of self-stigma
Self-stigma of patients perceived by their caregivers | 1 day during the scheduled consultation in the infectious diseases department of the Gabriel Montpied University Hospital in Clermont-Ferrand
  Percentage of caregivers who perceive self-stigma and how they propose to their patients the way to surpass themselves

CONTACTS AND LOCATIONS:
Overall Officials: Christine JACOMET, Dr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (43):
- France (41):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Chu Angers, Angers
  - CH Annecy Genevois, Annecy
  - Chru Besancon, Besançon
  - CHRU Brest, Brest
  - CH Cholet, Cholet
  - Hopital Antoine Beclere, Clamart
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Chu Dijon, Dijon
  - Hopital Raymond Poincaré, Garches
  - CHD Vendrée, La Roche-sur-Yon
  - Groupe Hospitalier de La rochelle-Ré-Aunis, La Rochelle
  - CH de Versailles, Le Chesnay
  - Hopital Bicetre Aphp, Le Kremlin-Bicêtre
  - Ch Le Mans, Le Mans
  - Centre Hospitalier Bretagne Sud, Lorient
  - CHU LYON, Lyon
  - CISIH, Marseille
  - Ch Montlucon, Montluçon
  - CH Morlaix, Morlaix
  - CH Moulins-Yzeure, Moulins
  - CHU de Mulhouse, Mulhouse
  - Chu Nantes, Nantes
  - CHU NICE, Nice
  - CH NIORT, Niort
  - CH Orléans, Orléans
  - Hopitel Necker, Paris
  - CH Perpignan, Perpignan
  - Chu Poissy, Poissy
  - CHU Poitiers, Poitiers
  - Centre Hospitalier Intercommunal de Cornouaille, Quimper
  - Pole Santé Publique - CH Laennec, Quimper
  - Chu Reims, Reims
  - CHU Nord, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - Hopital Tenon, Thenon
  - Chu Toulon, Toulon
  - Ch Valenciennes, Valenciennes
  - CHBA Vannes, Vannes
  - CH VICHY, Vichy
  - Hôpital Nord Ouest villefranche sur Saone, Villefranche-sur-Saône
- CHU Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe
- CHU Felix Guyon, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No